CLINICAL TRIAL: NCT01901666
Title: ASSESSMENT OF GH-IGF1 AXIS AND TO STUDY RESPONSE TO GH THERAPY IN CHILDREN WITH CML IN REMISSION HAVING GH DEFICIENCY
Brief Title: Assessment Of Gh-Igf-1 Axis In Children With Chronic Myelogenous Leukemia (CML) In Remission
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, dr anuradha aggarwal, senior resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GH-IGF-1 AXIS AND CML
Record Dates: First submitted 2013-06-29; First posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Myelogenous Leukemia; Short Stature
Keywords: growth hormone, Chronic Myelogenous Leukemia, Imatinib,serum IGF-1
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Dwarfism | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Growth hormone deficient group (Experimental): 0.3mg/kg/week GH in seven divided doses will be given subcutaneously for one year.
  Interventions: Drug: Growth Hormone

INTERVENTIONS:
Drug: Growth Hormone — All GH deficient patients with bone age <14 years will be treated with GH therapy for one year.Serum IGF-1 will be measured 4weekly and GH dose will be titrated till S.IGF-1 is in mid-normal range and then after every 3 months.
  Growth parameters will be assessed after every 3 months.Serum T4, TSH will be done after every 3 months. Patients will be monitored for any side effects of GH therapy
  Other Names: Recombinant human growth hormone

SUMMARY:
CML is a myeloproliferative disorder defined by the presence of the Philadelphia chromosome, which arises from the reciprocal translocation of genes on chromosomes 9 and 22.It is rare in childhood and accounts for 2-3% of all leukemias in childhood.

BCR-ABL gene on Philadelphia chromosome results in a 210kd fused BCR-ABL protein with constitutive tyrosine kinase activity, and subsequent activation of cytoplasmic and nuclear signal transduction pathways including STAT, RAS, JUN, MYC, and phosphatidylinositol-3 kinase. The ultimate result of such activation is the myeloid proliferation and differentiation and suppressed apoptosis.

Children present with a higher WBC count, otherwise presentation is nearly identical to adults. Current treatment include tyrosine kinase inhibitors (TKI) and allogeneic stem cell transplant (SCT).Imatinibmesylate inhibits the tyrosine kinase (TK) activity of BCR-ABL1 and several related TKs, including c-kit and the platelet-derived growth factor receptor (PDGFR). Development of tyrosine kinase inhibitor (TKI) therapy has revolutionizedtreatment of CML. Imatinib or second generation TKIs (dasatinib or nilotinib) have become standard front-line therapy forchildren and adults with CML and are also important componentsof therapy for Ph+ acute lymphoblastic leukemia (ALL).

TKIs are administered orally and cause a number of side effects including fatigue, hypertension, rash, impaired wound healing, myelosuppression, and diarrhea . The overall toxicity of TKIs, while less life-threatening than conventional cytotoxic chemotherapy, nevertheless is common, and may require dose reduction.Recently, proposed endocrine-related side effects of these agents include alterations in thyroid function, bone metabolism, linear growth, gonadal function, fetal development, glucose metabolism and adrenal function.

Growth impairment is one of the major adverse effect of long-term imatinib treatment in children with CML. Multiple case reports have demonstrated growth retardation in children onimatinib.Imatinibmesylate inhibits the TK activity of BCR-ABL1 and several related TKs, including c-kit and theplatelet-derived growth factor receptor (PDGFR). It isthe inhibition of TK activity at the non-BCR-ABL sites that couldbe the likely cause for the adverse effect on growth. Severalstudies in adults have suggested that inhibition of c-kit,c-fms, and PDGF receptors results in modulation of bone metabolism. Other reports are focusing on disturbance of the growth hormone (GH) axis as a mechanism for growth impairment. Receptor and non receptor TK is expressed at multiple levels in GH-IGF-1 axis including GHRH-R, GH-R and IGF-1R. Inhibition of TKs with TKI, at any one of these level, might result in growth impairment.

Various studies are available to show that Imainib therapy may cause short stature in children on prolonged treatment but exact mechanism by which this occurs is still not clear. Further, no treatment modality has been tried so far, for short stature in these children.

So, the purpose of this study is to study GH-IGF1 axis in these children and to administer GH therapy to GH deficienct children in remission.

DETAILED DESCRIPTION:
AIMS AND OBJECTIVES:

* To study GH-IGF1 axis in children with CML having short stature following Imatinib therapy.
* To administer growth hormone therapy to children with CML on Imatinib in remission having GH deficiency.

STUDY DESIGN: It is an interventional, non-randomized study. STUDY GROUP: one NUMBER OF PATIENTS: 20

ELIGIBILITY CRITERIA:

CML patients on Imatinib therapy for more than 6 months and in remission will be included in the study if there is:

* Severe short stature (height SDS <-3 SD)
* Severe growth deceleration (height velocity SDS <-2 SD over 12 months)
* Height <-2 SD and height velocity <-1.0 SD over 12 months
* Height <-1.5 SD and height velocity <-1.5 SD over 2 years

EXCLUSION CRITERIA:

* Patients with coexisting systemic illness (e.g. kidney disease, liver disease, celiac disease)
* Patients of CML not receiving Imatinib therapy as prescribed. (e.g. poor compliance)

MATERIALS AND METHODS:

Once eligibility criteria are confirmed, after having written informed consent, following parameters will be assessed:

* Chronological age
* Height
* Height for age
* Height SDS
* Target height
* Body proportion
* Weight
* Weight for age

Following investigations will be done in all patients:

* Complete blood count with peripheral smear.
* Liver function tests
* Renal function tests
* Calcium, phosphate, ALP, albumin.
* Fasting Blood glucose
* Thyroid function tests (T4, and TSH)
* Serum Cortisol
* Serum Prolactin
* Serum Follicular stimulating hormone (FSH) and Luteinizing hormone (LH)
* Serum Testosterone
* Serum Estrogen
* Serum IgA anti-tTG antibodies
* Serum IGF-1.
* Serum IGFBP-3.
* X-Ray of left hand and wrist
* MRI Brain focussing pituitary hypothalamic region. Two dynamic growth hormone provocation,GHRH + Arginine andGlucagon tests will be performed in all patients having no other cause for short stature.Minimum gap of one week will be kept between the two GHstimulationtests.Priming will be done prior to each GH stimulation test. IGF-1 generation test will be performed in all patients.Minimum gap of one week will be kept betweenGH stimulation and IGF-1 generation test.

X-ray of left hand and wrist for bone age and sexual maturity rating (SMR) by Tanners scale will be performed for all patients. All GH deficient patients with bone age <14 years will be treated with GH therapy for one year. 0.3mg/kg/week GH in seven divided doses will be given subcutaneously. Serum IGF-1 will be measured 4weekly and GH dose will be titrated till S.IGF-1 is in mid-normal range and then after every 3 months.

Patients will be monitored for any side effects of GH therapy Growth parameters, Serum T4, TSH and complete blood count will be assessed after every 3 months.Cytogenetic and molecular remission will be assessed before and after completion of GH therapy.

ELIGIBILITY:
Inclusion Criteria:

CML patients on Imatinib therapy for more than 6 months and in remission will be included in the study if there is

1. severe short stature (height SDS <-3 SD)
2. severe growth deceleration (height velocity <-2 SD over 12 months)
3. Height <-2 SD and height velocity <-1.0 SD over 12 months
4. Height <-1.5 SD and height velocity <-1.5 SD over 2 years

Exclusion Criteria:

1. Patients with coexisting systemic illness(e.g. kidney disease, liver disease, celiac disease).
2. Patients of CML not receiving Imatinib therapy as prescribed (poor compliance).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To know whether patients of CML who are faltering on growth after imatinib therapy are GH deficient or having GH resistance by performing GH provocation tests and IGF-1 generation test. | 30 months
  Growth impairment is one of the major adverse effect of long-term imatinib treatment in children with CML. Receptor and non receptor TK is expressed at multiple levels in GH-IGF-1 axis including GHRH-R, GH-R and IGF-1R. Inhibition of TKs with TKI, at any one of these level, might result in growth impairment.Various studies are available to show that Imainib therapy may cause short stature in children on prolonged treatment but exact mechanism by which this occurs is still not clear.So, the purpose of this study is to study GH-IGF1 axis in these children

SECONDARY OUTCOMES:
To administer growth hormone therapy to children with CML on Imatinib in remission having GH deficiency and to measure IGF-1 levels, gain in height and height velocity on GH therapy. | 12 months
  Disturbance of the growth hormone (GH) axis has been shown as one of the mechanism for growth impairment. But, no treatment modality has been tried so far for short stature in these children. So, one of the outcome measure will be to study gain in height after administeration of GH therapy to these GH deficient children.

CONTACTS AND LOCATIONS:
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Uttarakhand, India